CLINICAL TRIAL: NCT04492722
Title: A Phase 2b Randomised, Double-Blind, Placebo-Controlled, Multi-Centre, Dose-Ranging Study of AZD5718 in Participants With Proteinuric Chronic Kidney Disease
Brief Title: A Study to Evaluate the Safety and Efficacy of AZD5718 in Participants With Proteinuric Chronic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to terminate the study early due to lack of efficacy. There were no safety concerns related to the study.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry); Emerald Clinical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7551C00001; 2020-002263-54 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease
Keywords: Nephrology; Chronic kidney disease; Proteinuria; Diabetic kidney disease; Diabetes mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria; Diabetic Nephropathies; Diabetes Mellitus | interventions — AZD5718; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No member of the study team at AstraZeneca, or representative, personnel at study centres, or any CRO handling data will have access to the randomization scheme prior to unblinding for the primary analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZD5718 Dose 1 + Dapagliflozin 10 mg (Experimental): Participants will receive once daily oral dose 1 of AZD5718 for 12 weeks, thereafter add-on therapy of 10 mg dapagliflozin for 8 weeks.
  Interventions: Drug: AZD5718; Drug: Dapagliflozin 10 mg
- AZD5718 Dose 2 + Dapagliflozin 10 mg (Experimental): Participants will receive once daily oral dose 2 of AZD5718 for 12 weeks, thereafter add-on therapy of 10 mg dapagliflozin for 8 weeks.
  Interventions: Drug: AZD5718; Drug: Dapagliflozin 10 mg
- AZD5718 Dose 3 + Dapagliflozin 10 mg (Experimental): Participants will receive once daily oral dose 3 of AZD5718 for 12 weeks, thereafter add-on therapy of 10 mg dapagliflozin for 8 weeks.
  Interventions: Drug: AZD5718; Drug: Dapagliflozin 10 mg
- Placebo + Dapagliflozin 10 mg (Placebo Comparator): Participants will receive once daily oral dose of placebo matched to AZD5718 for 12 weeks, thereafter add-on therapy of 10 mg dapagliflozin for 8 weeks.
  Interventions: Drug: Dapagliflozin 10 mg; Drug: Placebo

INTERVENTIONS:
Drug: AZD5718 — Participants will receive once daily oral dose of AZD5718 as per the arms they are randomised, and will continue until Week 20.
  Arms: AZD5718 Dose 1 + Dapagliflozin 10 mg; AZD5718 Dose 2 + Dapagliflozin 10 mg; AZD5718 Dose 3 + Dapagliflozin 10 mg
Drug: Dapagliflozin 10 mg — Participants will receive once daily oral dose of 10 mg dapagliflozin for 8 weeks as an add-on therapy.
Drug: Placebo — Participants will receive once daily oral dose of placebo matched to AZD5718, and will continue until Week 20.
  Arms: Placebo + Dapagliflozin 10 mg

SUMMARY:
The purpose of the study is to evaluate the dose-response efficacy, safety, and pharmacokinetics (PK) of AZD5718 in participants with proteinuric chronic kidney disease.

DETAILED DESCRIPTION:
The study will be conducted in approximately 118 study centers across 12 countries. The overall study period will be around 28 weeks. Approximately 632 participants comprising of 67% diabetic kidney disease (DKD) and 33% non-DKD participants will be enrolled. After a screening period of up to 4 weeks, the participants will be randomised in a 1:1:1:1 ratio to receive one of the doses of AZD5718 and/or placebo for the first 12 weeks (Day 85 [treatment period 1]), with an add-on therapy of 8 weeks of dapagliflozin for all participants from Week 12 to 20 (Day 85 to 141 [treatment period 2]). Only participants still taking their assigned treatment from treatment period 1 will progress to treatment period 2. Any participant with urine albumin to creatinine ratio (ACR) < 30 mg/g at Week 12 will be excluded from treatment period 2. The eligibility check to enter treatment period 2 will be done at Visit 7 (Week 12) using the last available urine ACR result. The final analysis will be done after all participants have completed follow-up period of up to 4 weeks. The expected total study duration, including the Screening Period, for each participant will be at least 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent form.
* Male or female adults, >= 18 years of age at study entry.
* For participants who haven't reached the age of maturity according to local regulations in their country, a written informed consent should be obtained from the participant and participants legally acceptable representative.
* Body weight within 50-150 kg and body mass index within the range 18 to 45 kg/m^2.
* Participants with proteinuric CKD defined as:

  * eGFR 20 - 75 mL/min/1.73m^2 based on Chronic Kidney Disease Epidemiology Collaboration equation at Screening Visit 1.
  * Albuminuria defined as 200 -5000 mg albumin/g creatinine based on the geometric mean of the replicated measurements using 3 sequential first morning void urine at Visit 2.
  * Participants with diagnosis of Type 2 Diabetes Mellitus (DM) [for DKD sub-group only].
* Females of non-childbearing potential must have been surgically sterilized or be postmenopausal, and all female participants must have a negative pregnancy test at screening and prior to study drug administration.
* Male participants must be surgically sterile or agree to use highly effective contraceptives. Non-sterilized male participants who are sexually active with a female partner of childbearing potential must use a male condom with spermicide from Day 1 to 3 months after the last dose of the study drug. Approved/Certified measurements in Japan are as Vasectomy, tubal occlusion, intrauterine device (provided coils are copper banded), levonorgestrel intrauterine system (eg, Mirena®). These measurements are acceptable forms of highly effective birth control in Japan. Not Approved/Certified measurements in Japan are as: Cerazette® (desogestrel) pills, medroxyprogesterone injections (eg, Depo-Provera®), etonogestrel implants (eg, Implanon®, Norplan®), normal and low dose combined oral pills, norelgestromin/ethinylestradiol transdermal system (eg, Evra® Patch), intravaginal device (eg, NuvaRing®).
* Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of samples for optional exploratory genetic research.
* Participants should have: a) stable blood pressure (BP [BP <= 150/100 mmHg at Visit 1, and 3]); b)stable dose of angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blockers (ARB) for at least 4 weeks prior to Screening Visit 1; c) participants who have been unable to tolerate ACEi or ARB therapy may be enrolled.
* Participants must have been on a stable dose for at least 4 weeks prior to Screening Visit 1, who have been on additional antihypertensives (including diuretics); on treatment with drugs with potential to influence albuminuria eg., non-steroidal anti-inflammatory drug; on renin inhibitor or an aldosterone antagonist in combination with an ACEi or an ARB.
* Participants on Sodium-glucose co-transporter-2 inhibitors (SGLT2i) or Glucagon-like peptide-1 receptor agonist (GLP1-RA) treatment, the participants must have been on a stable dose for at least 4 weeks prior to randomization visit.

Exclusion Criteria:

* Participants with recent positive hepatitis B or hepatitis C.
* Diagnosis of polycystic kidney disease or anatomical causes of CKD.
* Diagnosis of Type 1 DM.
* Participants with severe hepatic impairment (Child-Pugh class C).
* Abnormal laboratory findings at Screening Visit 1.
* Any of the following concomitant conditions or diseases at Screening Visit 1:

  1. History of QT prolongation associated with other medications that required discontinuation of that medication, and congenital long QT syndrome.
  2. Acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass grafting within 6 months.
  3. High degree atrioventricular block II-III, sinus node dysfunction.
  4. Stroke within 3 months, heart failure, and anticipated dialysis or renal transplantation within 1 year.
  5. Any other condition or clinically relevant abnormal findings in physical examination, laboratory results or ECG during screening period.
  6. History of substance dependence or a positive screen for drugs or alcohol abuse. Alcohol and drug screening to be completed for all participants locally with laboratory kits provided by the central laboratory.
* Participant who had severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated), and/or had a confirmed case of COVID-19 within 4 weeks of Screening Visit 1.
* Ongoing use of any biologic drug and/or small molecule targeting the immune system.
* Any serum creatinine-altering drugs within 1 month prior to Screening Visit 1.
* Treatment with any concomitant medications known to be associated with Torsades de Pointes or potent inducers/inhibitors of cytochrome P450 3A4 within 4 weeks of Visit 3 (Randomization).
* Treatment with zileuton, cilastatin (dipeptidase-1 [DPEP1] inhibitor), or leukotriene receptor antagonists (eg, montelukast) within 4 weeks of Screening Visit 1.
* Treatment with simvastatin, lovastatin, and atorvastatin at doses > 40 mg per day within 1 month prior to Screening Visit 1.
* Concurrent enrollment in another clinical study involving an investigational treatment or drug or participation in a device study within 3 months prior to Screening Visit 1.
* Participants with a known hypersensitivity to AZD5718 or any of the excipients of the product. Participants with a known hypersensitivity to dapagliflozin or any of the excipients of the product.
* Donation of blood or significant blood loss in excess of 500 mL within 3 months prior to Day 1 (or > 1200 mL in the year prior to Day 1).
* Plasma donation within 60 days prior to Day 1.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study center).
* Judgement by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
* For women only - currently pregnant (a negative serum pregnancy test is required at Screening Visit 1 and urine pregnancy test at Day 1 [Visit 3]) or breast-feeding.
* An employee, or close relative of an employee, of AstraZeneca, the Contract Research Organisation, or the study site, regardless of the employee's role.
* Participants who are legally institutionalized.
* Participants working night shifts, and who cannot avoid strenuous manual labour during the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiddo J. L. Heerspink, Principal Investigator — Department of Clinical Pharmacy and Pharmacology University Medical Centre Groningen
Locations (88):
- United States (22):
  - Research Site, Canoga Park, California
  - Research Site, La Mesa, California
  - Research Site, San Carlos, California
  - Research Site, San Francisco, California
  - Research Site, Victorville, California
  - Research Site, Denver, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Roseville, Michigan
  - Research Site, Hazelwood, Missouri
  - Research Site, Fresh Meadows, New York
  - Research Site, Great Neck, New York
  - Research Site, Jamaica, New York
  - Research Site, Blue Ash, Ohio
  - Research Site, East Providence, Rhode Island
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Schertz, Texas
- Argentina (5):
  - Research Site, Bahía Blanca
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Junín
  - Research Site, Mar del Plata
- Brazil (8):
  - Research Site, Belém
  - Research Site, Brasília
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Meireles
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São Paulo
- Germany (4):
  - Research Site, Aschaffenburg
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Trier
- Hungary (5):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szentes
  - Research Site, Szigetvár
- Israel (5):
  - Research Site, Afula
  - Research Site, Ashdod
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
- Japan (15):
  - Research Site, Ageo
  - Research Site, Asahikawa-shi
  - Research Site, Chiba
  - Research Site, Hiroshima
  - Research Site, Kasugai-shi
  - Research Site, Kitakyushu
  - Research Site, Koga-shi
  - Research Site, Kyoto
  - Research Site, Mito
  - Research Site, Morioka
  - Research Site, Osaka
  - Research Site, Sashima-gun
  - Research Site, Shizuoka
  - Research Site, Toride-shi
  - Research Site, Yokohama
- Malaysia (6):
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Malacca
  - Research Site, Seremban
  - Research Site, Seri Manjung
  - Research Site, Sibu
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Oświęcim
  - Research Site, Rzeszów
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
- Ukraine (8):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Heerspink HJL, Law G, Psachoulia K, Connolly K, Whatling C, Ericsson H, Knochel J, Lindstedt EL, MacPhee I. Design of FLAIR: a Phase 2b Study of the 5-Lipoxygenase Activating Protein Inhibitor AZD5718 in Patients With Proteinuric CKD. Kidney Int Rep. 2021 Aug 27;6(11):2803-2810. doi: 10.1016/j.ekir.2021.08.018. eCollection 2021 Nov. PMID 34805632
- See also: Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7551C00001&attachmentIdentifier=d8fc6532-dec8-43e7-937b-828cf4d0d085&fileName=CSP.pdf&versionIdentifier=
- See also: Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7551C00001&attachmentIdentifier=18780c46-89ba-4175-b893-33b0b39ce0bf&fileName=SAP.pdf&versionIdentifier=
- See also: Clinical Study Results Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7551C00001&attachmentIdentifier=817aeaff-7ef5-4bdc-8cd2-858d351426a0&fileName=CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 01 October 2020 to 06 September 2022. The study was terminated early on 01 July 2022 due to lack of efficacy.
Pre-assignment Details: The screening period was for 4 weeks. Participants who met all the inclusion and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- AZD5718 Dose 1 + Dapagliflozin 10 mg: Participants received once daily oral dose of AZD5718 Dose 1 for 12 weeks, and thereafter an add-on therapy of 10 mg dapagliflozin for 8 weeks.
- AZD5718 Dose 2 + Dapagliflozin 10 mg: Participants received once daily oral dose of AZD5718 Dose 2 for 12 weeks, and thereafter an add-on therapy of 10 mg dapagliflozin for 8 weeks.
- AZD5718 Dose 3 + Dapagliflozin 10 mg: Participants received once daily oral dose of AZD5718 Dose 3 for 12 weeks, and thereafter an add-on therapy of 10 mg dapagliflozin for 8 weeks.
- Placebo + Dapagliflozin 10 mg: Participants received once daily oral dose of placebo matched to AZD5718 for 12 weeks, thereafter add-on therapy of 10 mg dapagliflozin for 8 weeks.
Period: Overall Study
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg | Placebo + Dapagliflozin 10 mg
Started | 154 | 153 | 153 | 153
Completed | 72 | 82 | 82 | 82
Not Completed | 82 | 71 | 71 | 71
Not completed — Adverse Event | 7 | 2 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 6 | 6 | 0 | 3
Not completed — Development of Study Specific Withdrawal Criteria | 3 | 1 | 2 | 2
Not completed — Due to Covid-19 pandemic | 7 | 3 | 7 | 6
Not completed — Failure to meet randomisation criteria | 2 | 3 | 4 | 2
Not completed — Early termination from the study | 54 | 51 | 50 | 50
Not completed — Missing | 3 | 0 | 0 | 5
Not completed — Participants who did not receive treatment | 0 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomised and received any study treatment were included in the Full Analysis Set (FAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg | Placebo + Dapagliflozin 10 mg | Total
Number analyzed (Participants) | 154 | 152 | 149 | 153 | 608
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (10.70) | 63.7 (10.63) | 65.1 (9.39) | 64.3 (10.71) | 64.5 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 53 | 45 | 53 | 208
  Male | 97 | 99 | 104 | 100 | 400
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 37 | 28 | 32 | 129
  Not Hispanic or Latino | 122 | 115 | 121 | 121 | 479
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 54 | 55 | 56 | 52 | 217
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 20 | 16 | 15 | 15 | 66
  White | 68 | 73 | 67 | 77 | 285
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 8 | 11 | 9 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Reduction of Urine Albumin to Creatinine Ratio (ACR) to Week 20
Description: The dose response effect of AZD5718 on urine ACR at 20 weeks was evaluated. Values less than 1 indicate improvement from baseline.
Time Frame: Week 1 (Baseline) to Week 20
Population: Per-protocol analysis set consisted of all participants who received the additional treatment with dapagliflozin post-Week 12 and who did not violate the terms of the protocol in a way that could affect the primary efficacy endpoint significantly.
Measure: Geometric Mean (95% Confidence Interval); unit: milligram/gram (mg/g)
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg | Placebo + Dapagliflozin 10 mg
Number analyzed (Participants) | 69 | 67 | 75 | 76
milligram/gram (mg/g) | 0.79 [0.69 to 0.90] | 0.81 [0.70 to 0.92] | 0.77 [0.67 to 0.87] | 0.84 [0.73 to 0.95]

2. Secondary Outcome: Change From Baseline in Reduction of Urine ACR to Week 12
Description: The dose response effect of AZD5718 on urine ACR at 12 weeks was evaluated. Values less than 1 indicate improvement from baseline.
Time Frame: Week 1 (Baseline) to Week 12
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg | Placebo + Dapagliflozin 10 mg
Number analyzed (Participants) | 99 | 97 | 101 | 104
mg/g | 0.94 [0.84 to 1.04] | 1.03 [0.92 to 1.15] | 0.96 [0.86 to 1.06] | 1.10 [0.99 to 1.22]

3. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: The safety and tolerability profile of AZD5718 treatment was assessed
Time Frame: From Screening (Week -4 to 0) to Week 24
Population: All participants who were randomised and received any study treatment. Participants were evaluated according to the actual treatment they received. If a participant had received a different treatment dose than randomised throughout the study, they would have been analysed according to the treated dose, not the randomisation dose.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg | Placebo + Dapagliflozin 10 mg
Number analyzed (Participants) | 154 | 152 | 149 | 153
Participants
  Any AE | 82 | 81 | 104 | 80
  Any AE with outcome = death | 0 | 0 | 0 | 1
  Any SAE (including events with outcome = death) | 12 | 8 | 11 | 6
  Any AE leading to discontinuation of study treatment | 12 | 2 | 3 | 6
  Any AE leading to dose interruption | 7 | 6 | 5 | 10
  Any AE leading to withdrawal from study | 7 | 0 | 1 | 1
  Any AE possibly related to study treatment as assessed by investigator | 14 | 12 | 8 | 14

4. Secondary Outcome: Change From Baseline in 24-hours Mean Systolic Blood Pressure to Week 12
Description: The effect of AZD5718 on ambulatory blood pressure was assessed
Time Frame: Week 1 (Baseline) to Week 12
Population: All participants in the Full Analysis Population who had valid Ambulatory Blood Pressure data for change from baseline analyses.
Measure: Mean (Standard Deviation); unit: millimeter mercury (mm Hg)
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg | Placebo + Dapagliflozin 10 mg
Number analyzed (Participants) | 69 | 78 | 70 | 85
millimeter mercury (mm Hg) | -2.06 (10.782) | 1.56 (11.407) | -1.83 (9.986) | 3.76 (11.779)

5. Secondary Outcome: Plasma Concentrations of AZD5718
Description: The PK of AZD5718 after repeated oral dosing for 20 weeks was evaluated
Time Frame: From Week 2 to Week 20
Population: All participants in the Full Analysis Population who have at least one detectable AZD5718 plasma concentration measurement post-treatment. The Pharmacokinetic Population was used for all PK analyses. Here "n" is the number of participants included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg
Number analyzed (Participants) | 88 | 91 | 96
nanomoles per liter (nmol/L)
  Week 2 (pre-dose) | 4.771 (113.047) | 12.181 (116.038) | 37.346 (138.565)
  Week 4 (pre-dose): number analyzed (Participants) | 83 | 84 | 93
  Week 4 (pre-dose) | 3.975 (85.449) | 11.207 (111.951) | 37.525 (127.660)
  Week 8 (pre-dose): number analyzed (Participants) | 72 | 76 | 81
  Week 8 (pre-dose) | 3.947 (77.097) | 11.579 (113.404) | 35.903 (116.207)
  Week 12 (pre-dose): number analyzed (Participants) | 70 | 69 | 75
  Week 12 (pre-dose) | 4.107 (79.068) | 11.041 (81.967) | 33.568 (127.405)
  Week 16 (pre-dose): number analyzed (Participants) | 54 | 54 | 59
  Week 16 (pre-dose) | 4.115 (76.378) | 10.006 (97.216) | 35.662 (130.148)
  Week 20 (pre-dose): number analyzed (Participants) | 45 | 47 | 51
  Week 20 (pre-dose) | 3.813 (65.605) | 10.200 (122.277) | 33.063 (100.320)
  Week 4 (post-dose, 1-2 hours): number analyzed (Participants) | 23 | 27 | 24
  Week 4 (post-dose, 1-2 hours) | 16.321 (115.673) | 71.279 (128.551) | 340.794 (147.394)
  Week 4 (post-dose, 2-5 hours): number analyzed (Participants) | 22 | 28 | 23
  Week 4 (post-dose, 2-5 hours) | 18.376 (77.409) | 86.464 (103.733) | 464.721 (79.567)
  Week 4 (post-dose, 5-8 hours): number analyzed (Participants) | 21 | 28 | 23
  Week 4 (post-dose, 5-8 hours) | 16.713 (65.648) | 76.834 (59.503) | 343.531 (90.628)
  Week 4 (post dose, 8-12 hours): number analyzed (Participants) | 21 | 28 | 23
  Week 4 (post dose, 8-12 hours) | 14.434 (52.414) | 53.706 (68.160) | 234.913 (97.174)

6. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) to Week 12
Description: The effect of AZD5718 on renal function was evaluated
Time Frame: Week 1 (Baseline), Week 2, Week 4, Week 8, and Week 12
Population: Per-protocol analysis set consisted of all participants who received the additional treatment with dapagliflozin post-Week 12.
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73m^2
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg | Placebo + Dapagliflozin 10 mg
Number analyzed (Participants) | 100 | 101 | 105 | 106
milliliter/minute/1.73m^2
  Week 2: number analyzed (Participants) | 100 | 100 | 105 | 106
  Week 2 | -0.470 (6.3936) | -0.140 (5.2801) | -0.429 (5.7175) | 0.547 (5.7124)
  Week 4: number analyzed (Participants) | 98 | 100 | 104 | 103
  Week 4 | -0.735 (6.5764) | 0.140 (5.2628) | -0.817 (6.1986) | 0.058 (6.3583)
  Week 8: number analyzed (Participants) | 100 | 101 | 104 | 103
  Week 8 | -0.760 (6.0304) | -0.535 (5.8865) | -1.144 (6.5142) | -0.068 (5.3729)
  Week 12: number analyzed (Participants) | 98 | 94 | 99 | 101
  Week 12 | -0.612 (6.2138) | -1.149 (6.1783) | -0.394 (6.4678) | -0.257 (6.4508)

ADVERSE EVENTS:
Time Frame: From Screening (Week -4 to 0) to Week 24
Arm/Group | AZD5718 Dose 1 + Dapagliflozin 10 mg | AZD5718 Dose 2 + Dapagliflozin 10 mg | AZD5718 Dose 3 + Dapagliflozin 10 mg | Placebo + Dapagliflozin 10 mg
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/152 | 0/149 | 1/153
Serious Adverse Events (participants affected / at risk) | 12/154 | 8/152 | 11/149 | 6/153
Other Adverse Events (participants affected / at risk) | 16/154 | 8/152 | 9/149 | 8/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD5718 Dose 1 + Dapagliflozin 10 mg (N=154) | AZD5718 Dose 2 + Dapagliflozin 10 mg (N=152) | AZD5718 Dose 3 + Dapagliflozin 10 mg (N=149) | Placebo + Dapagliflozin 10 mg (N=153)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pituitary apoplexy (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD5718 Dose 1 + Dapagliflozin 10 mg (N=154) | AZD5718 Dose 2 + Dapagliflozin 10 mg (N=152) | AZD5718 Dose 3 + Dapagliflozin 10 mg (N=149) | Placebo + Dapagliflozin 10 mg (N=153)
Urinary tract infection (Infections and infestations) | 8 (8) | 8 (8) | 1 (2) | 6 (6) — The Number of Events was less than the Number of Affected Participants.
Glomerular filtration rate decreased (Investigations) | 8 (9) | 3 (3) | 5 (9) | 8 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (7) | 9 (9) | 6 (9)

LIMITATIONS AND CAVEATS:
Following study termination and reduced scope of the analysis, the PK analysis has not been performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca. Access to this document must be restricted to relevant parties.

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT04492722/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT04492722/SAP_001.pdf